CLINICAL TRIAL: NCT03859531
Title: Gastrointestinal Outcome Measures Before and After Orkambi Therapy in Cystic Fibrosis (CF) Patients Carrying the F508del Mutation on Both Alleles
Brief Title: Gastrointestinal Study at Orkambi Therapy in CF Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: Hadassah Medical Organization (Other); Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Principal Investigator, Isabelle de Monestrol, Director of Stockholm CF Center, Karolinska University Hospital
Other Study IDs: CF-GI-001
Record Dates: First submitted 2019-02-26; First posted 2019-03-01 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CF patients planned to receive Orkambi: CF patients carrying the F508del mutation on both alleles planned to receive Orkambi therapy

SUMMARY:
Ivacaftor caused a significance increase in weight in patients carrying the G551D mutation and the etiology of this has largely remained unknown but may be due to improved function of the gastrointestinal tract. The combination therapy of Orkambi has been recently approved for subjects with Cystic Fibrosis homozygous for F508del mutation. This provides an opportunity to examine if there are any improvements in gastrointestinal function. The investigators aim to investigate various aspects of gastrointestinal and pancreatic function before and 6 months after the commencement of Orkambi therapy.

DETAILED DESCRIPTION:
To examine the entire intestinal mucosa via capsule endoscopy before and 6 months after Orkambi therapy to ascertain if the inflammatory changes in the intestine have improved. A marker of intestinal inflammation measured in the stool, Calprotectin, will be examined before and 6 months after Orkambi treatment. The investigators hypothesize that the result will be reduced on therapy.

A marker of pancreatic exocrine function, pancreatic elastase, will be examined before and 6 months after therapy to examine if the result has increased indicating improvement of exocrine pancreatic function

Study Population All subjects with CF homozygous for the F508del mutation in Sweden eligible for Orkambi therapy, i.e. above 12 years of age, in total 145 patients in Sweden of which 60 are taken care of at Stockholm CF Center; the investigators aim to examine 20 patients.

Study Duration The duration will be 6 months for each patient.

ELIGIBILITY:
Inclusion Criteria:

* CF patients F508del homozygote
* >12 years of age
* eligible for Orkambi therapy.

Exclusion Criteria:

* Patients who the patency capsule does not pass within 48 hrs
* FEV1<30%
* Pregnancy and breastfeeding women
* Liver function blood tests (AST, ALT, Gamma-GT, ALP) >3 xULN
* Bilirubin >2 xULN
* AST or ALT alone >5 xULN
* Previous lung transplant

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CF patients, F508del homozygote, >12 years of age, eligible and planned for Orkambi therapy in Clinical routine.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-02-27 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Concentration of fecal calprotectin | Change from baseline at 6 months after commencing treatment with Orkambi
  Is a marker of intestinal inflammation measured in the stool
Concentration of fecal elastase-1 | Change from baseline at 6 months after commencing treatment with Orkambi
  Is a test of pancreatic function measured in the stool.
Change in small bowel capsule endoscopy (SBCE) | Change from baseline at 6 months after commencing treatment with Orkambi
  The method of SBCE has been well established as a descriptive diagnostic tool for intestinal inflammation and has been used as an outcome measure in clinical trials. Erythema, petechiae, mucosal erosions and ulcerations will be assessed according to the Maiden criteria

SECONDARY OUTCOMES:
Change in CRP | Change from baseline at 6 months after commencing treatment with Orkambi
  Inflammatory marker, unit mg/L.
Change in sedimentation rate | Change from baseline at 6 months after commencing treatment with Orkambi
  Inflammatory marker, unit mm.
Concentration of serum electrophoresis. | Change from baseline, 6 months after commencing treatment with Orkambi
  Inflammatory markers: alpha-1-antitrypsin, haptoglobin, orosomucoid, immunoglobulin A, M and G.
Change in liver function tests | Change from baseline at 6 months after commencing treatment with Orkambi
  ALT, AST, ALP, gamma-GT. Unit: mikrokat/L
Change in bilirubin | Change from baseline at 6 months after commencing treatment with Orkambi
  Bilirubin. Unit: mikromol/L

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle de Monestrol, MD PhD, Principal Investigator — Stockholm CF Center
Locations (1):
- Stockholm CF Center, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Because this would expose the patients too much

REFERENCES:
- [Background] Borowitz D, Lubarsky B, Wilschanski M, Munck A, Gelfond D, Bodewes F, Schwarzenberg SJ. Nutritional Status Improved in Cystic Fibrosis Patients with the G551D Mutation After Treatment with Ivacaftor. Dig Dis Sci. 2016 Jan;61(1):198-207. doi: 10.1007/s10620-015-3834-2. Epub 2015 Aug 7. PMID 26250833
- [Background] Wainwright CE, Elborn JS, Ramsey BW. Lumacaftor-Ivacaftor in Patients with Cystic Fibrosis Homozygous for Phe508del CFTR. N Engl J Med. 2015 Oct 29;373(18):1783-4. doi: 10.1056/NEJMc1510466. No abstract available. PMID 26510034
- [Background] Werlin SL, Benuri-Silbiger I, Kerem E, Adler SN, Goldin E, Zimmerman J, Malka N, Cohen L, Armoni S, Yatzkan-Israelit Y, Bergwerk A, Aviram M, Bentur L, Mussaffi H, Bjarnasson I, Wilschanski M. Evidence of intestinal inflammation in patients with cystic fibrosis. J Pediatr Gastroenterol Nutr. 2010 Sep;51(3):304-8. doi: 10.1097/MPG.0b013e3181d1b013. PMID 20512061

DOCUMENTS (1):
  • Study Protocol (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/31/NCT03859531/Prot_000.pdf